CLINICAL TRIAL: NCT03854123
Title: Multiple Sclerosis in the Elderly: Epidemiology, Clinical and MRI Characteristics
Acronym: OLDMUS
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Observatoire Français de la sclérose en plaques (OFSEP) (Unknown); Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2014/02
Record Dates: First submitted 2018-04-05; First posted 2019-02-26 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Multiple Sclerosis
Keywords: Geriatric population; EDMUS; OFSEP
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Old MS patients: 75 to 77 years old MS patients whose disease began at 65 years old or earlier will be retrieved from the "Observatoire français de la sclérose en plaques" (OFSEP).

SUMMARY:
Little is known about old MS patients. In a previous work, systematic search in Bordeaux, Strasbourg and Dijon university hospital regional MS center databases European Database for Multiple Sclerosis (EDMUS) retrieved 2% of 75 years old or older Multiple Sclerosis (MS) patients in the 3 databases. Data analysis showed that MS may switch off in the very old patients with mild progression and very few relapses. The project is to continue this preliminary work and extend it with a systematic study of MS in the elderly.

The scientific aims: To add new insights into long lasting MS natural history in the growing population of elderly patients with MS.

DETAILED DESCRIPTION:
75 to 77 years old MS patients whose disease began at 65 years old or earlier will be retrieved from the "Observatoire français de la sclérose en plaques" (OFSEP) which includes more than 50 000 MS patients in France. Accuracy of these patients' data from 65 to 75 years old will be thereafter checked and completed in 3 French MS centers: Lyon, Rennes and Bordeaux, participating to this database directly from the patients' clinical files. From these 3 MS centers around 150 MS patients from 75 to 77 years old are expected to be analysed on site.

The data wich will be retrieved for these patients are: irreversible disability status scale progression, relapses, Magnetic Resonance Imaging (MRI) data, CSF data, Lublin classification of type of MS, McDonald 2005 and 2010 criteria, date and age at beginning of progression, characteristics and modality of relapses and clinical impairment at the beginning of the disease, treatments used, treatment failures and side effects, co morbidity, Barthel index, EuroQol-5D (EQ-5D), cognitive impairment (SDMT test), social life data and socio economic data. To the investigator's knowledge this will be the first systematic description of very old MS patients with data on long term natural history of MS and characteristics in this population of elderly MS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with McDonald 2001, 2005 or 2010 criteria of multiple sclerosis 75 to 77 years old MS patients at the time of inclusion
* Patients whose beginning of MS was before 65 years old or 65 years old
* Patients who signed OFSEP 's consent

Exclusion Criteria:

* Patients whose clinical data cannot be entered or for whom too much clinical data are missing
* Alive patients older than 77 years or younger than 75 years the day of the inclusion in the study
* Patients died before 65 years old

Ages: 75 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 75 to 77 years old MS patients whose disease began at 65 years old or earlier will be retrieved from the "Observatoire français de la sclérose en plaques" which includes more than 50 000 MS patients in France.
Sampling Method: Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
Evaluation of MS evolution with disability progression (irreversible Disability Status Scale) in 75 to 77 years Old MS Patients from the age of 65 years-old to present time | At inclusion (day 0)
  Time to reach the irreversible Kurtzke disability status scale (DSS) score 4, 6 and 7

SECONDARY OUTCOMES:
Frequency of clinical relapses in 75 years Old or Older MS Patients from the age of 65 years-old to present time | At inclusion (day 0)
Description of the clinical characteristics at 75 years Old | At inclusion (day 0)
  Clinical conversion to secondary progressive MS date
Description of the Cerebral MRI at 75 years Old | At inclusion (day 0)
  Number of lesions on T2 sequence if <9, number of new T2 lesions, Number of Gadolinium enhancing lesions, T1-Hypointense Lesions (T1 Black Holes), MRI Barkhof Criteria and number of periventricular lesions if <3,
Description of the paraclinical characteristics at 75 years Old | At inclusion (day 0)
  Distance walked (with or without help)
Description of the paraclinical characteristics at 75 years Old | At inclusion (day 0)
  Barthel index
Socio-demographic data | At inclusion (day 0)
  sex
Socio-demographic data | At inclusion (day 0)
  age
Socio-demographic data | At inclusion (day 0)
  department of residence
Description of the treatments at 75 years Old | At inclusion (day 0)
  Treatments of multiple sclerosis
Description of the treatments at 75 years Old | At inclusion (day 0)
  Failures treatments of multiple sclerosis
Description of the treatments at 75 years Old | At inclusion (day 0)
  Side effects of treatments and other concomitant treatments
Measure of health-related quality of life at 75 years Old | At inclusion (day 0)
  EQ-5D Instruments
Evaluation of cognitive functions at 75 years Old | At inclusion (day 0)
  Symbol digit modalities test (SDMT) test

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe OUALLET, MD, PhD, Principal Investigator — CHU de Bodeaux; Sandra VUKUSIC, Prof., Study Chair — Observatoire Français de la sclérose en plaques (OFSEP)
Locations (3):
- France (3):
  - CHU de Bordeaux - Pellegrin - service de neurologie, Bordeaux
  - Hôpital neurologique - Pierre Wertheimer, Bron
  - CHU de Rennes - service de neurologie, Rennes